CLINICAL TRIAL: NCT03495037
Title: Preventing Cognitive and Functional Decline Among Seniors at Risk: A Community-Based Randomized Trial
Brief Title: Preventing Cognitive and Functional Decline Among Seniors at Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Dr. Deirdre Dawson, Senior Scientist, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REB1738
Record Dates: First submitted 2018-02-22; First posted 2018-04-11 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Subjective Cognitive Decline
Keywords: Age-related cognitive changes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real World Strategy Training (Experimental): Group intervention including education and strategy training to manage everyday functional difficulties.
  Interventions: Behavioral: Real World Strategy Training
- Psychosocial Education (Active Comparator): Group sessions including education on brain health.
  Interventions: Behavioral: Psychosocial Education

INTERVENTIONS:
Behavioral: Real World Strategy Training — The key features of the protocol are: i. Participants are actively engaged in selecting their treatment goals. The research clinician will work with the participants to identify five specific, measurable real-world goals using a standardized semi-structured interview, the Canadian Occupational Performance Measure. Three of these will be training goals, two will not be trained but evaluated post-intervention for evidence of generalization and transfer to non-trained tasks; ii. A global problem solving approach is used (Goal- Plan- Do- Check). Participants are guided by the trainer to apply this strategy to their goals.
  Other Names: Adopted Cognitive Orientation to Occupational Performance
  Arms: Real World Strategy Training
Behavioral: Psychosocial Education — The active comparator uses an information-based format and is designed to engage participants without providing any specific training techniques or strategies. During weekly sessions, participants will receive factual information on brain structure and function, age-related cognitive changes, and general brain health issues and will spend time doing non-specific cognitive exercises including crossword and Sodoku puzzles. Homework will consist of reading assignments related to the session topics.
  Arms: Psychosocial Education

SUMMARY:
This study evaluates the efficacy of Real-World Strategy Training (RWST) compared to a psycho-education workshop for improving everyday life performance in older adults with subjective cognitive decline (SCD). Participants will be randomly assigned to receive one of these approaches.

DETAILED DESCRIPTION:
Evidence suggests that 25-50% of community-dwelling older adults report SCD and that these individuals have an elevated risk for developing Mild Cognitive Impairment and/or dementia. Many of these individuals report difficulties with complex activities of daily living.

RWST aims to reduce these difficulties in everyday life by providing a meta-cognitive training approach that compensates for age-related executive changes. The approach is provided within the context of individually identified everyday-life difficulties.

The psycho-education approach is a Brain-Health Workshop supplemented by intellectually stimulating activities such as doing Sudoku and/or word searches. This approach provides information people may use to inform health behaviour changes.

ELIGIBILITY:
Inclusion Criteria:

* Have subjective cognitive complaints
* Be fluent in written and spoken English
* Able to self-identify areas of their everyday lives in which they would like to improve.

Exclusion Criteria:

* Diagnosis of neurological conditions (e.g. dementia, mild cognitive impairment, Parkinson's)
* Presence of severe depression
* Presence of substance abuse
* History of hospitalization for psychiatric reasons

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in improved performance (measured as total number of untrained goals improved to criterion) on the Canadian Occupational Performance Measure (COPM) immediately post-intervention. | Changes from baseline to post-intervention at 10 weeks.
  The COPM is a standardized semi-structure interview in which participants identify everyday life difficulties (defined as things they need to or want to do). These issues are converted to goals with performance rated on a 10-point Likert-type scale. Goals considered improved to criterion are those that have a 2 or more points increase on ratings.

SECONDARY OUTCOMES:
Improved performance on the Canadian Occupational Performance Measure (COPM) measured at three and six months post-intervention. | Three and six months post-intervention.
  See primary outcome.
Improved satisfaction with performance on trained and untrained goals identified using the COPM. | 10 weeks after baseline (after intervention), 3 months post-intervention, 6 months post-intervention.
  Satisfaction with performance is measured on a 10-point Likert type scale using the COPM.
Improved performance on the Multiple Errands Test (MET). | 10 weeks after baseline (after intervention), 3 months post-intervention, 6 months post-intervention.nths post-intervention.
  The MET is an ecologically valid, performance measure being used to determine if strategies learned in RWST are transferred to novel contexts. Best performance is achieved through completing all tasks (n=12) without breaking any rules (n=9).
Change in health-related Quality of Life | Baseline, 10 weeks, 3 months post-intervention, 6 months post-intervention.
  Health-related quality of life will be measured using the SF-36.
Improved performance on neuropsychological measures of executive function. | Baseline, 10 weeks, 3 months post-intervention, 6 months post-intervention.
  Changes in executive function are anticipated as meta-cognitive strategy training targets the executive control system. These will be measured using the Delis-Kaplan Executive Function System.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Dawson, PhD, Principal Investigator — Rotman Research Institute, Baycrest Health Sciences
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada